CLINICAL TRIAL: NCT00526045
Title: A Phase I Dose Escalation, Multi-center, Open-label Study of AUY922 Administered IV on a Once Weekly Schedule in Adult Patients With Advanced Solid Malignancies Including Phase II Expansion Arms in Patients With Either HER2 Positive or ER Positive Locally Advanced or Metastatic Breast Cancer.
Brief Title: Phase I-II Study to Determine the Maximum Tolerated Dose (MTD) of AUY922 in Advanced Solid Malignancies, and Efficacy in HER2+ or ER+ Locally Advanced or Metastatic Breast Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAUY922A2101; 2006-002766-20 (EudraCT Number)
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2013-05

CONDITIONS: Breast Cancer; Hematologic Neoplasms
Keywords: AUY922; Solid tumors; Breast Cancer; Phase I/II; Advanced Solid malignancies (Phase I); Breast Cancer ( Phase II ); HER2+; ER+; HSP90
MeSH Terms: conditions — Breast Neoplasms; Hematologic Neoplasms | interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide

ARMS (3):
- Escalation (Experimental)
  Interventions: Drug: AUY922 2 mg/m2
- HER2 Positive (Experimental)
  Interventions: Drug: AUY922 2 mg/m2
- ER+ breast cancer (Experimental)
  Interventions: Drug: AUY922 2 mg/m2

INTERVENTIONS:
Drug: AUY922 2 mg/m2

SUMMARY:
This is a phase I/II, open-label, multicenter study of AUY922 administered intravenously in patients with advanced solid malignancies to determine the maximum tolerated dose. Phase II expansion arms will investigate efficacy in patients with either HER2 positive or ER positive locally advanced or metastatic breast cancer. Additional patients with advanced solid malignancies will also be investigated in a separate expansion arm. Safety, pharmacokinetics and pharmacodynamics will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Dose-escalation and MTD dose expansion arm: Patients with histologically confirmed, advanced malignant solid tumors whose disease has progressed on standard therapy or for whom no standard therapy exists.

   Breast cancer phase II expansion arms only:
   1. Females patients with HER2 positive non-operable locally advanced or metastatic breast cancer must have:

      * History of trastuzumab resistance, defined as either local or systemic disease progression on treatment with at least 8 weeks of a trastuzumab containing regimen.
      * Received up to 3 prior anti HER2 based regimens (i.e. trastuzumab and/or lapatinib in combination with other agents) for metastatic disease
      * Patients who develop metastases while receiving adjuvant or neo-adjuvant trastuzumab are eligible.

      HER2 positive patients, tumor/s must demonstrate HER2 over-expression based on either:
      * Immunohistochemistry (IHC) at the 3+ level, or
      * IHC 2+ confirmed by fluorescence in-situ hybridization (FISH). Tumors tested by FISH must be positive by the specific FISH assay for the amplification of HER2.
   2. Female patients with ER positive non-operable locally advanced or metastatic breast cancer patients who received standard sequence lines of endocrine therapy and whose disease has progressed on at least one and up to 3 lines of endocrine and/or cytotoxic therapy for advanced disease.
2. All patients must have at least one measurable lesion as defined by RECIST. Irradiated lesions are only evaluable for disease progression.
3. All patients must have progressive disease before entering the study
4. Age ≥ 18 years.
5. World Health Organization (WHO) Performance Status of ≤ 2.
6. Life expectancy of ≥ 12 weeks.
7. Absolute Neutrophil Count (ANC) 1.5 x 109/L; hemoglobin (Hgb) 9 g/dl; platelets (plt) 100 x 109/L; potassium, calcium, magnesium and phosphorus within normal limits or correctable with supplements; AST/SGOT and ALT/SGPT ≤ 2.5 x Upper Limit of Normal (ULN) or ≤ 5.0 x ULN if liver metastases are present; serum bilirubin 1.5 x ULN; serum albumin > 2.5g/dl and serum creatinine 1.5 x ULN or 24-hour clearance 50 ml/min

Exclusion criteria:

1. Patients with CNS metastasis which are:

   * Symptomatic or
   * Require treatment for symptom control and/or
   * Growing

   Note: patients without clinical signs or symptoms of CNS involvement are not required to have a CT/MRI of the brain
2. Prior treatment with any HSP90 or HDAC inhibitor compound.
3. Patient who received systemic anti-cancer treatment prior to the first dose of AUY922 within the following time frames:

   * Chemotherapy within 4 weeks
   * Radiotherapy within 4 weeks
   * Palliative radiotherapy: within 2 weeks
   * Trastuzumab treatment within 4 weeks
   * Nitrosoureas, mitomycin and monoclonal antibodies (except trastuzumab): within 6 weeks
   * Any continuous-dosing (i.e. daily dosing, every-other-day dosing, Monday- Wednesday-Friday dosing, weekly etc) of systemic anticancer treatment for which the recovery period is not known, or investigational drugs (i.e. targeted agents) within a duration of ≤ 5 half lives of the agent and their active metabolites (if any)
4. Patients who have not recovered from side effects of previous systemic anticancer therapy to less than grade 2 CTCAE prior to the first dose.
5. Pregnant or lactating women.
6. Cardia exclusion criteria:

   * History (or family history) of long QT syndrome.
   * Mean QTc ≥ 450 msec on screening ECG
   * History of clinically manifest ischemic heart disease including myocardial infarction, stable or unstable angina, coronary arteriography or cardiac stress testing/imaging with findings consistent with coronary occlusion or infarction, ≤ 6 months prior to study start.
   * History of heart failure or left ventricular (LV) dysfunction (LVEF ≤ 45%) by MUGA or ECHO
7. Known diagnosis of HIV infection (HIV testing is not mandatory).
8. Acute or chronic liver disease, acute or chronic renal disease or other concurrent severe and/or uncontrolled medical conditions (e.g. uncontrolled diabetes, active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol.
9. Cardiac exclusion criteria:

Mean QTc ≥ 450 msec on screening ECG and clinically significant ECG abnormalities including one or more of the following: left bundle branch block (LBBB), right bundle branch block (RBBB) with left anterior hemiblock (LAHB). ST segment elevations or depressions > 1mm, or 2nd (Mobitz II) or 3rd degree AV block; clinically significant ECG abnormalities including one or more of the following: left bundle branch block (LBBB), right bundle branch block (RBBB) with left anterior hemiblock (LAHB). ST segment elevations or depressions > 1mm, or 2nd (Mobitz II) or 3rd degree AV block.

History (or family history) of long QT syndrome, heart failure or left ventricular (LV) dysfunction (LVEF ≤ 45%) by MUGA or ECHO, history of clinically manifest ischemic heart disease including myocardial infarction, stable or unstable angina, coronary arteriography or cardiac stress testing/imaging with findings consistent with coronary occlusion or infarction, ≤ 6 months prior to study start; history or presence of atrial fibrillation, atrial flutter or ventricular arrhythmias including ventricular tachycardia or Torsades de Pointes.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2007-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The safe dose of AUY922 when administered once a week | 54 weeks (MTD determination)

SECONDARY OUTCOMES:
Efficacy of AUY922 administered once a week | Baseline, and every 2 cycles (time to document tumor progression)
Pharmacokinetics of AUY922 and Pharmacodynamics by PET response, blood and tumor biomarkers at baseline and post-AUY922 | Baseline and every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- United States (7):
  - UCLA/ University of California Los Angeles UCLA, Los Angeles, California
  - Georgia Health Sciences University Med College of GA, Augusta, Georgia
  - Dana Farber Cancer Institute StudyCoordinator:CAUY922A2101, Boston, Massachusetts
  - Washington University School Of Medicine-Siteman Cancer Ctr Dept. of Siteman Cancer Ctr., St Louis, Missouri
  - Nevada Cancer Institute Clinical Trials Office, Las Vegas, Nevada
  - MD Anderson Cancer Center/University of Texas Thoractic Head/Neck Med.Onc(2), Houston, Texas
  - Cancer Therapy & Research Center / UT Health Science Center InstituteForDrugDevelopment(3), San Antonio, Texas
- Novartis Investigative Site, Groningen, Netherlands
- Novartis Investigative Site, Bellinzona, Switzerland
- Novartis Investigative Site, Sutton, United Kingdom

REFERENCES:
- See also: Resutls for CAUY922A2101 on the Novartis clinical trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=8324